CLINICAL TRIAL: NCT01427530
Title: Local Field Potentials Recorded From Deep Brain Stimulating Electrodes Implanted for the Treatment of Parkinson's Disease
Brief Title: Local Field Potentials Recorded From Deep Brain Stimulating (DBS) Electrodes
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0511M77707
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Parkinson's Disease
Keywords: brain activity; implanted with DBS electrodes
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation

SUMMARY:
This study will be recording and evaluating brain activity from Deep Brain Stimulating (DBS) electrodes in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Surgical Candidate for DBS implantation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients undergoing DBS implantation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
recording and evaluating brain activity from Deep Brain Stimulating (DBS) electrodes in patients with Parkinson's disease. | At baseline
  recording and evaluating brain activity from Deep Brain Stimulating (DBS) electrodes in patients with Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Abosch, MD, Principal Investigator — University of Minnesota
Locations (1):
- Department of Neurosurgery, University of Minnesota, Minneapolis, Minnesota, United States